CLINICAL TRIAL: NCT01123005
Title: Imaging and Biomarkers of Hypoxia in Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Logistical
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Billy W. Loo Jr., Associate Professor of Radiation Oncology, Stanford University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-15039; VAR0032 (Other: OnCore)
Record Dates: First submitted 2009-07-27; First posted 2010-05-13 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — Magnetic Resonance Spectroscopy; carbogen; Dichloroacetic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Carbogen arm (Experimental)
  Interventions: Procedure: PET Scan; Drug: EF5; Drug: Carbogen
- DCA arm (Experimental)
  Interventions: Procedure: PET Scan; Drug: EF5; Drug: Dichloroacetate

INTERVENTIONS:
Procedure: PET Scan — radiation calculated per patient
  Other Names: positron emission tomography
Drug: EF5 — 10 mCi, IV
  Other Names: NSC-684681
Drug: Carbogen — Calculated per patient
  Other Names: Meduna's Mixture
  Arms: Carbogen arm
Drug: Dichloroacetate
  Other Names: DCA
  Arms: DCA arm

SUMMARY:
Hypoxia, meaning a lack of oxygen, has been associated strongly with a wide range of human cancers. Hypoxia occurs when tumor growth exceeds the ability of blood vessels to supply the tumor with oxygenated blood. It is currently understood that hypoxic tumors are more aggressive. Current methods for measuring hypoxia include invasive procedures such as tissue biopsy, or insertion of an electrode into the tumor. EF5-PET may be a non-invasive way to measure tumor hypoxia.

DETAILED DESCRIPTION:
To establish PET imaging with the tracer EF5 as an accurate and reliable method for measuring the oxygen content of a tumor and to establish the measurement of secreted markers in blood as an accurate and reliable method for measuring the oxygen content of a tumor.

ELIGIBILITY:
INCLUSION CRITERIA

* Any solid tumor malignancies of any stage meeting all of the following criteria: Minimum tumor dimension is at least 1 cm (to ensure it is above the detection threshold of PET imaging). Examples include but are not limited to: locally advanced squamous cell carcinoma of the head and neck to be treated by either initial surgery or primary chemoradiotherapy; inoperable non-small cell lung cancer or pancreatic carcinoma to be treated with stereotactic radiotherapy, which may be biopsied again at the time of percutaneous needle delivery of implanted fiducial markers.
* Patients with newly diagnosed malignancies should not have initiated treatment for their disease before participating in this study. Patients with recurrent or second malignancies may have had prior therapy as appropriate for their disease, but should have completed all prior treatment at least 30 days before participation in this study and should not have initiated new treatment for the current problem.
* Greater than or equal to eighteen years of age.
* Sufficiently healthy to tolerate all study procedures.
* Organ and marrow function sufficient to undergo planned therapy.
* Ability to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA

• Pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2010-12; Primary Completion 2015-08-21 (Actual); Study Completion 2015-08-21 (Actual)

PRIMARY OUTCOMES:
18F-EF5 uptake (tumor: blood ratio) before and after carbogen breathing for a subset of subjects. | 1-5 days
18F-EF5 uptake (tumor: blood ratio) before and after administration of DCA for a subset of subjects. | 1-5 days

SECONDARY OUTCOMES:
Levels of secreted hypoxia markers in plasma. | 1-5 days
Hypoxia gene and protein expression scores in patients undergoing biopsy or surgical resection. | 1-5 days

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Billy W. Loo Jr. M.D. Ph.D., Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No